## Janssen Research & Development \*

# Statistical Analysis Plan Week 24 (Primary) and Week 48 (Final) Analysis

A Phase 2, Open-label, Single-arm, Multicenter Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Switching to RPV Plus Other ARVs in HIV-1-infected Children (Aged 2 to <12 years) who are Virologically Suppressed

Protocol TMC278HTX2002; Phase 2

**Edurant®/TMC278(rilpivirine)** 

**Status:** Approved

**Date:** 27 March 2023

**Prepared by:** Janssen Research & Development, a division of Janssen Pharmaceutica NV

**Document No.:** EDMS-ERI-196339540

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

## **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TAB | ABLE OF CONTENTS2 | |
|---|---|---|
| AME | ENDMENT HISTORY | 4 |
| ABB | BREVIATIONS | 4 |
| 1 | INTRODUCTION | G |
| 1.<br>1.1. | Trial Objectives | |
| 1.1. | | |
| 1.2. | Trial Endpoints | |
| 1.3. | Trial Design | |
| 1.4. | Statistical Hypotheses for Trial Objectives | |
| 1.5.<br>1.6. | | |
| 1.7. | Randomization and Blinding | |
| 2. | GENERAL ANALYSIS DEFINITIONS | 8 |
| 2.1. | Analysis Phases. | |
| 2.2. | Visit Windows | |
| 2.3. | Pooling Algorithm for Analysis Centers | |
| 2.4. | Analysis Sets | |
| 2.4.1. | | |
| 2.4.2. | • | |
| 2.5. | Definition of Subgroups | |
| 2.6. | Study Day and Relative Day | |
| 2.7. | Baseline | |
| 2.8. | Imputation Rules for Missing AE Date/Time of Onset/Resolution | |
| 3. | INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW | 11 |
| 4. | SUBJECT INFORMATION | |
| 4.1. | Demographics and Baseline Characteristics | |
| 4.2. | Disposition Information | |
| 4.3. | Treatment Adherence | |
| 4.4. | Extent of Exposure | |
| 4.4.1. | | |
| 4.5. | Protocol Deviations | |
| 4.6. | Prior and Concomitant Medications | 15 |
| 5. | EFFICACY | |
| 5.1. | Analysis Specifications | |
| 5.1.1. | C | |
| 5.1.2. | $\epsilon$ | |
| 5.2. | Efficacy Endpoints | |
| 5.2.1. | | |
| 5.2.2. | • | |
| 5.3.<br>5.3.1. | Other Efficacy Variables | |
| <b>6.</b> 6.1. | SAFETY | |
| 6.2. | | |
| 6.3. | Clinical Laboratory Tests Vital Signs and Physical Examination Findings | |
| 6.4. | Electrocardiogram | |
| 7. | PHARMACOLOGY | |
| 7.1. | Population Pharmacokinetics | |
| / . 1 . | 1 operation 1 narmacokinetics | 20 |

# Statistical Analysis Plan TMC278HTX2002 (W24 &W48 Analysis)

| Pharma<br>7.2. | cokinetic/Pharmacodynamic Relationships | 26<br>27 |
|---|---|---|
| REFER | RENCES | . 28 |
| ATTAC | CHMENTS | . 29 |
| ATTAC | CHMENT 1: DAIDS GRADING TABLE | . 29 |
| ATTAC | CHMENT 2: BLOOD PRESSURE LEVELS BY AGE AND HEIGHT PERCENTILES | 34 |
| | CHMENT 3: STAGE-3-DEFINING OPPORTUNISTIC ILLNESSES IN HIV INFECTION | |

## **AMENDMENT HISTORY**

NA

#### **ABBREVIATIONS**

17-OH 17-hydroxyprogesteron

3TC lamivudine ABC abacavir

ACTH adrenocorticotropic hormone

ADaM Analysis Data Model AE Adverse Events

AESI Adverse Events of Special Interest

ALT alanine transaminase ART antiretroviral therapy

ARV antiretroviral

AST aspartate transaminase

ATC Anatomic and Therapeutic Chemical

AUC area under the curve

AZT zidovudine

BMI Body Mass Index

CD4 cluster of differentiation 4

CDC Centers for Disease Control and Prevention

CI Confidence Interval

cm centimeter

CRF Case Report Form DAIDS Division of AIDS

DHEAS dehydroepiandrosterone-sulfate
DPS Data Presentation Specifications

ECG electrocardiogram

eGFR estimated glomerular filtration rate

EOI event of interest
FAS Full Analysis Set
FC Fold Change

FDA Food and Drug Administration

FPI First Patient In

FSH Follicle-stimulating hormone

FTC Emtricitabine FU Follow Up

HIV-RNA Human immunodeficiency virus Ribonucleic Acid

HR Heart Rate

IDMC Independent Data Monitoring Committee
ICH International Conference on Harmonization

IVRS interactive voice response system

kg Kilogram

LH luteinizing hormone

LOCF Last Observation Carried Forward

NC Non Completer

MedDRA Medical Dictionary for Regulatory Activities

mL millilitre

MTCT Mother to Child Transmission

NAP Not Applicable

N(t)RTI nucleoside/nucleotide reverse transcriptase inhibitors

nmol nanomol

PBMC peripheral blood mononuclear cell

PD Pharmacodynamic
PK Pharmacokinetic(s)
q.d. quaque die (one a day)
QTc corrected QT interval

QTcB Bazett's square-root corrected QT QTcF Fridericia's square-root corrected QT

RPV Rilpivirine

SAE Serious Adverse Events
SAP Statistical Analysis Plan
SD Standard Deviation

SDTM Study Data Tabulation Model

SE Standard Error

SI International System of Units TLF Tables, Listings and Figures

TLOVR Time to Loss of Virologic Response

WHO-DD World Health Organization-Drug Dictionary

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables, and statistical methods for the Week 24 (primary) and Week 48 (final) analysis of safety and efficacy (antiviral activity) of the study TMC278HTX2002 based on the protocol version 16.0 dated 22 February 2021 (Amendment 3).

## 1.1. Trial Objectives

## Primary Objectives:

- To evaluate the steady-state Pharmacokinetic (PK) of rilpivirine (RPV) and determine the appropriate dose of RPV in combination with other antiretrovirals (ARVs) in participants aged ≥2 to <12 years with a body weight of <25kg.
- To evaluate the safety and tolerability of RPV in combination with other ARVs in participants aged ≥2 to <12 years over a 24-week treatment period.

## Secondary Objectives:

- To evaluate the safety and tolerability of RPV in combination with other ARVs over a 48-week treatment period.
- To evaluate the efficacy of RPV in combination with other ARVs over a 24- and 48-week treatment period.
- To evaluate population PK and PK/pharmacodynamic (PD) relationships for safety and efficacy of RPV in combination with other ARVs.
- To assess resistance in case of loss of virologic response to RPV in combination with other ARVs.
- To evaluate treatment adherence to RPV in combination with other ARVs over a 24- and 48-week treatment period.

## **Exploratory Objectives:**

- To assess the palatability of the 2.5-mg tablet formulation of RPV, if applicable.
- To assess the swallowability of the 25-mg tablet formulation of RPV, if applicable.
- To assess archived viral resistance, if feasible depending on available blood volume.

## 1.2. Trial Endpoints

## **Primary Endpoints:**

- Area under the plasma concentration-time curve from time of administration up to 24 hours post-dose of RPV, as derived from the intensive PK assessments.
- Incidence of grade 3/4 adverse events (AEs), serious adverse events (SAEs), Human Immunodeficiency Virus (HIV)-related events (including acquired immune deficiency syndrome [AIDS]-defining illnesses and Stage-3-defining Opportunistic Illnesses in HIV Infection), and AEs leading to discontinuation of study intervention through 24 weeks of study treatment.

## Secondary Endpoints:

- Incidence and severity of AEs/HIV-related events and their relatedness to RPV through 24 and 48 weeks of study treatment.

- Change from baseline over time and shift in toxicity grades/abnormalities versus reference for clinical laboratory parameters, electrocardiogram (ECG) parameters, vital signs, and physical examination through 24 and 48 weeks of study treatment.
- Proportion of participants with HIV-1 RNA <50/400 and ≥50/400 copies/mL using the Food and Drug Administration (FDA) Snapshot approach through 24 and 48 weeks of study treatment.
- Immunologic changes, measured by CD4+ cell count (absolute and percentage relative to total lymphocytes), through 24 and 48 weeks of study treatment.
- Pharmacokinetic parameters of RPV (other than area under the plasma concentration-time curve [AUC]), as derived from the intensive PK assessments.
- Pharmacokinetic parameters of RPV, as derived by population PK modeling, through 24 and 48 weeks of study treatment.
- Viral genotype at the time of virologic failure through 24 and 48 weeks of study treatment.
- Treatment adherence, as assessed by the Pediatric European Network for the Treatment of AIDS (PENTA) adherence questionnaire and by study intervention accountability, through 24 and 48 weeks of study treatment.

#### **Exploratory Endpoints:**

- Responses to the palatability questionnaire after 2 weeks of study treatment.
- Responses to the swallowability questionnaire after 2 weeks of study treatment.
- Mutations in HIV-1 DNA or in HIV-1 RNA, as assessed by retrospective peripheral blood mononuclear cell (PBMC)- or plasma-based analyses, through 24 and 48 weeks of study treatment.

## 1.3. Trial Design

This is a Phase 2, open-label, single-arm, multicenter, interventional study in HIV-1-infected participants (boys and girls) aged  $\geq 2$  to  $\leq 12$  years with a body weight of at least 10kg to evaluate the PK, safety, tolerability, and efficacy of switching to RPV once daily in combination with other, investigator-selected ARVs.

For more details refer section 4 of the study protocol.

# 1.4. Statistical Hypotheses for Trial Objectives

No formal hypothesis will be tested.

## 1.5. Sample Size Justification

No formal sample size calculation was performed.

The sample size is based on overall regulatory requirements and the number of participants enrolled in Cohort 2 in study TMC278-C213: approximately 25 to 30 participants aged  $\geq$ 2 to <12 years will be recruited in the current study.

For more details refer section 9.2 of the study protocol.

## 1.6. Randomization and Blinding

## Randomization

As this was a single arm trial, no randomization procedures were applicable.

## **Blinding**

Since this was an open label trial, blinding procedures were not applicable.

## 1.7. Changes to planned analyses

**NAP** 

#### 2. GENERAL ANALYSIS DEFINITIONS

## 2.1. Analysis Phases.

Table 1 – Trial Phases

| Trial phase | Start date | End date |
|---|---|---|
| Screening | Date of signing the informed consent | Start date of Treatment phase - 1 day |
| Treatment | Date of the first intake of RPV | If the participant <i>died during the study</i> intervention phase: min (date of last RPV+ 7 days; date of death) If the participant permanently stopped the trial medication: minimum of: ■ date of last RPV intake + 7 days, if missing, max (early withdrawal visit date; discontinuation date) + 7 days ■ date of last contact [For W24 analysis only] If the participant is still in the trial: cut-off date for the analysis, ie. LPW24 visit date |
| Follow-up (not<br>defined when<br>derived End<br>date is before<br>Start date of this<br>phase) | End date of the Treatment phase + 1 day | If the participant <i>died</i> : date of death Otherwise: date of last contact (or cut-off date for the analysis, if still in follow-up period) |

If the date of first intake of the study medication is missing, this should be substituted by the baseline visit date.

## 2.2. Visit Windows

As participants do not always adhere to the protocol visit schedule, the following rules are applied to assign actual visits to analysis visits. Listed below are the visit windows and the target days for each visit. The reference day is Study Day 1. If a participant has 2 or more actual visits in one visit window, the visit closest to the target day will be used as the protocol visit for that visit window. The other additional visit(s) will not be used in the summaries or analyses, but they can be used for determination of clinically important endpoints. If 2 actual visits are equidistant from the target day within a visit window, the later visit is used.

All assignments will be made in chronological order. Once a visit date is assigned to a visit window, it will no longer be used for a later time point except for the endpoint. Listed below (Table 2) are the visit windows and the target days for each visit defined in the protocol.

Table 2 – Visit Windows

| Parameter | Analysis<br>Period | Scheduled<br>Visit Number | Time Interval (label on output) | Time Interval<br>(Day)** | Target Time<br>Point (Day) |
|---|---|---|---|---|---|
| Vital Signs* | Screening | 1 | Screening | <0 | -∞ |

| Parameter | Analysis<br>Period | Scheduled<br>Visit Number | Time Interval (label on output) | Time Interval (Day)** | Target Time<br>Point (Day) |
|---|---|---|---|---|---|
| | Baseline § | 2 | Baseline | [ <b>-</b> ∞, 1] | ≤1 |
| | | 3 | Week 2 | [2,21] | 15 |
| | | 4 | Week 4 | [22, 42] | 29 |
| | | 5 | Week 8 | [43, 70] | 57 |
| | | 6 | Week 12 | [71, 98] | 85 |
| | T | 7 | Week 16 | [99, 140] | 113 |
| | Treatment | 8 | Week 24 | [141, 196] | 169 |
| | | 9 | Week 32 | [197, 252] | 225 |
| | | 10 | Week 40 | [253, 308] | 281 |
| | | 11 | Week 48 | [309, 378] | 337 |
| | Follow-up | 12 | Post-treatment | [Start FU phase, | (3x7) + 1 = 22 |
| | | | Follow-up | $\infty$ ] | after Start FU |
| | | | | | phase |

<sup>\*</sup>Vital Signs used as an example refer parameter which data collected on each protocol schedule visit

## 2.3. Pooling Algorithm for Analysis Centers

NAP.

## 2.4. Analysis Sets

# 2.4.1. All Enrolled Analysis Set

The all enrolled analysis set includes all participants who were not screen failures.

## 2.4.2. Full Analysis Set (FAS)

The FAS includes all participants who have taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen.

The FAS will be used as primary and only population for all analyses.

## 2.5. Definition of Subgroups

All results will be presented by age group (2-<6 years; 6-<12 years) as well as overall across whole study population.

In addition, the following subgroups defined:

## Efficacy:

- CD4<sup>+</sup> count at baseline (< 350, 350 < 500, 500 < 750,  $\geq$ 750 cells/ $\mu$ L) [Note: last 2 categories may be combined into 1]
- Background regimen (ie. ABACAVIR/LAMIVUDINE, Other)

<sup>\*\*</sup>Relative to Study Day 1

<sup>§</sup> Only the record prior to the first dose closest to target day 1 will be allocated to analysis time point 'Baseline'; all records prior to Day 1 that were not allocated to Baseline are assigned to 'Screening'.

 Adherence based on drug accountability (<80%, 80 - <95%, >=95%) cumulative up to Week 24/ Week 48

## Safety:

- Baseline body weight: <15 kg; 15 kg <20 kg; 20 <25 kg; at least 25 kg
- RPV dose (12.5mg, 15mg, 25mg)
- CD4<sup>+</sup> count at baseline (< 350, 350 < 500, 500 < 750,  $\geq$ 750 cells/ $\mu$ L) [Note: last 2 categories may be combined into 1]
- Background regimen (ie. ABACAVIR/LAMIVUDINE, Other)

# 2.6. Study Day and Relative Day

Study Day 1 or Day 1 refers to the start of the first study agent administration (date of first intake). All efficacy and safety assessments at all visits will be assigned a day relative to this date.

Study day or relative day for a visit is defined as:

Study Day = visit date - date of Day 1 + 1; if visit date  $\geq$  date of Day 1 (date of first study treatment (RPV) administration).

Study Day = visit date – date of Day 1; if visit date < date of Day 1 (date of first study treatment (RPV) administration).

There is no 'Day 0'

#### 2.7. Baseline

A baseline (or reference) value will be defined as the value of the last available assessment prior to the first study treatment (RPV) on Day 1.

If the baseline value is missing the last available screening value will be taken.

## 2.8. Imputation Rules for Missing AE Date/Time of Onset/Resolution

Partial AE onset dates will be imputed as follows:

• If the onset date of an adverse event is missing day only, it will be set to:

First day of the month that the AE occurred, if month/year of the onset of AE is different than the month/year of the study agent start

The day of study agent start, if the month/year of the onset of AE is the same as month/year of the study agent start date and month/year of the AE resolution date is different

The day of study agent start or day of AE resolution date, whichever is earliest, if month/year of the onset of AE and month/year of the study agent start date and month/year of the AE resolution date are same

• If the onset date of an adverse event is missing both day and month, it will be set to the earliest of:

January 1 of the year of onset, as long as this date is on or after the study agent start date. Month and day of the study agent start date, if this date is the same year that the AE occurred Last day of the year if the year of the AE onset is prior to the year of the study agent start date,

The AE resolution date.

Edurant®/TMC278(rilpivirine)

• Completely missing onset dates will not be imputed.

Partial AE resolution dates not marked as ongoing will be imputed as follows:

- If the resolution date of an adverse event is missing day only, it will be set to the earliest of the last day of the month of occurrence of resolution or the day of the date of death, if the death occurred in that month.
- If the resolution date of an adverse event is missing both day and month, it will be set to the earliest of December 31 of the year or the day and month of the date of death, if the death occurred in that year.
- Completely missing resolution dates will not be imputed.

AE onset/resolution dates with missing times will be imputed as follows:

- A missing time of onset of an adverse event will be set to the earlier of:
  - 00:01 as long as the onset date is after the study agent start date
  - The time of the study agent start if this is the same day the AE occurred.
- The missing time of resolution of an adverse event will be set to 23:59.

If a missing time is associated with a partial or missing date, the date will be imputed first prior to imputing the time.

## 3. INTERIM ANALYSIS AND DATA MONITORING COMMITTEE REVIEW

An Independent Data Monitoring Committee (IDMC) was installed to monitor pharmacokinetic, efficacy, and safety data, and to safeguard the participants in this trial.

Interim analyses were performed and presented to the IDMC at Week 4, at Week 12 when all participants reached Week 12 (or discontinued earlier) and primary analysis at Week 24 when all participants reached Week 24 (or discontinued earlier). The details of these analyses are described in the corresponding IDMC SAPs. The Week 48 (final) analysis when all participants have completed the trial up to Week 48 (or discontinued earlier) will be shared and discussed with the IDMC.

Further details are described in the IDMC charter.

#### 4. SUBJECT INFORMATION

The number of participants in FAS will be summarized and listed by age group (2-<6 years; 6-<12 years) and overall.

## 4.1. Demographics and Baseline Characteristics

Table 3 presents a list of the demographic variables that will be summarized.

Table 3: Demographic Variables

| Continuous Variables: | Summary Type |
|-------------------------------|----------------------------------|
| Age (years) | Descriptive statistics (N, mean, |
| Weight (kg) | standard deviation [SD], median, |
| Height (cm) | and range [minimum and |
| Body Mass Index (BMI) (kg/m2) | maximum]). |
| Categorical Variables | |

11

| Age ( $\ge 2$ - < 6years; $\ge 6$ - < 9years; $\ge 9$ - < 12years) | Frequency distribution with the |
|---|---|
| Weight (<25kg, ≥25kg) | number and percentage of |
| Sex (male, female) | participants in each category. |
| Childbearing Potential (Yes, No) | |
| Race <sup>a</sup> (American Indian or Alaska Native, Asian, Black or African | |
| American, Native Hawaiian or other Pacific Islander, White, Not allowed | |
| to ask per local regulations, Multiple) | |
| Ethnicity (Hispanic or Latino, not Hispanic or Latino, Not allowed to ask | |
| per local regulations) | |
| Country <sup>b</sup> | |

<sup>&</sup>lt;sup>a</sup> If multiple race categories are indicated, Race is recorded as 'Multiple'

Table 4 presents a list of the baseline disease characteristic variables that will be summarized.

**Table 4: Baseline Disease Characteristic Variables** 

| Continuous Variables: | Summary Type |
|---|---|
| CD4+ count (cells/μL) at Baseline | |
| CD4+ count (%) at Baseline | |
| HIV-1 viral load (copies/ml / log <sub>10</sub> copies/ml) at Baseline | |
| Duration of known HIV Infection (years): | |
| [date of first confirmed positive HIV-1 test – date of Day 1]/365.25 | Descriptive statistics (N, mean, |
| <i>Note</i> : provide duration in years; in case of incomplete date of first | standard deviation [SD], median, and |
| confirmed positive HIV test, impute with the 1st day of the month | range [minimum and maximum]). |
| and/or 1st month of the year in order to derive the duration. | |
| Categorical Variables | |
| HIV – 1 subtype (from historical report or PBMC) | |
| Hepatitis B/C co-infection status (Yes, No, NAV) | |
| Mode of HIV infection (Blood transfusion, Hemophilia-associated | |
| injections, Mother to Child transmission, Other) | Frequency distribution with the number and percentage of participants in each category. |
| Clinical stage of HIV infection at screening based on CD4+ count OR | |
| percentage of total lymphocytes | |
| CD4+ count at Baseline (< 350, 350 - < 500, 500 - <750, $\geq$ 750 cells/ $\mu$ L) | |
| HIV-1 viral load at Baseline (<50 copies/ml and ≥50 copies/ml) | |

## 4.2. Disposition Information

Screened participants and reason for screen failures will be summarized overall.

The number of participants in the following disposition categories will be summarized throughout the study by age group (2-<6 years; 6-<12 years) and overall.

For the All Enrolled Analysis Set:

- Participants enrolled
- Participants enrolled but not treated
- Participants treated with study treatment (FAS)

## and for FAS:

- Participants completing the study
- Participants who terminated study participation prematurely
- Reasons for termination of study

<sup>&</sup>lt;sup>b</sup> Summary will be detailed for sites in each country

#### 4.3. Treatment Adherence

Treatment adherence is defined based on drug accountability and based on the Study Adherence Questionnaire for Children and Teenagers / the Study Adherence Questionnaire for Caregivers (see Appendix 10 of the Clinical Trial Protocol).

The following parameters are derived cumulatively up to week 24 or week 48/last intake for discontinued participants as well as using all available data (Week 24 analysis only).

Treatment adherence will be summarized descriptively by age group (2-<6 years; 6-<12 years) and overall for the entire 24-Week and 48-Week treatment period.

## Drug Accountability:

Drug accountability (DA) can only be calculated at time points when all kits that have been dispensed before that time point have been returned – if DA cannot be derived (eg. cumulative up to week 24):

- impute with value based on next available time point for which a DA calculation can be done, eg. if cumulative DA up to week 24 cannot be derived, derive DA up to week 32; if not calculable, derive DA up to week 40 etc.;
- otherwise, use value based on closest preceding time point

Total Amount to be taken (in mg) =

 $\sum_{across\ RPV\ doses}$  (number of days on same RPV dose x strength in mg of RPV dose)

Number of days on same RPV dose is based on:

first and last RPV study medication intake date (if available) of the prescribed RPV dose
or, in case participant discontinued and last RPV study medication intake date is missing,
discontinuation date

Actual Total amount taken (in mg) =

 $\sum_{across\ RPV\ doses}$  ((number of tablets dispensed – number of tablets returned) x strength in mg of RPV tablet)

Level of adherence = (actual Total amount taken / Total amount to be taken) x 100%

Treatment adherence is defined as:

- adherent: the level of adherence is > 95%
- non-adherent: the level of adherence is  $\leq 95\%$

Additionally, following categories of level of adherence will be defined: -

- > 95%
- ]80%; 95%]
- [165%; 80%]
- [50%; 65%]
- $\le 50\%$

The numbers and percentages of participants by adherence category will be tabulated and descriptive statistics of adherence (%) will be shown.

Interruptions (for AEs) are not to be considered for the calculation of adherence, i.e. they will not be subtracted from the Total amount to be taken.

## **PENTA Questionnaires:**

Source for this adherence measure is the Study Adherence Questionnaire for Children and Teenagers (or, when completed by the caregiver, the Study Adherence Questionnaire for Caregivers), more specifically the following 2 questions:

- i. Report of missed doses in last 3 days (Question 8).
- ii. Report of missed doses over the last 2 weeks (Question 9).

If both child and a caregiver completed the questionnaire, the Child Questionnaire will be given precedence.

Results will be summarized for RPV and for the background regimen separately (regardless which ARVs are used) – in case questionnaire results for >1 ARV are reported concurrently, the worst outcome (eg. higher # doses missed for Q8) across these ARVs will be used in the analysis, and further as follows:

- i. Missed doses in last 3 days (Q8):
  - on a by visit basis (0, 1, 2, or 3 doses missed)
  - cumulatively, with the following categories and subcategories:
    - 1. never missed a dose
    - 2. missed not more than 1 dose
      - a. at most once
      - b. more than once
    - 3. missed 2 or more doses
      - a. at most once
      - b. more than once
- ii. Missed doses (Y/N) in last 2 weeks (Q9):
  - on a by visit basis (Y/N)
  - cumulatively, with the following categories and subcategories:
    - 1. never missed doses
    - 2. missed doses.
      - a. at most once
      - b. more than once

Treatment adherence, for both RPV and background regimen, is defined as:

- adherent: cumulatively, did not miss (2 or more) doses more than once (i.1., i.2.(a&b), i.3.a, ii.1, and ii.2.a)
- non-adherent: cumulatively, missed (2 or more) doses more than once (i.3.b or ii.2.b)

## 4.4. Extent of Exposure

The number and percentage of participants who receive RPV will be summarized by age group (2-<6 years; 6-<12 years) and overall.

Exposure is defined as the duration of RPV treatment. The duration is calculated as follows:

(date of last dose of RPV - date of first dose of RPV) + 1.

Note that this definition implies that drug interruptions are ignored in calculating exposure.

Descriptive statistics for RPV duration in weeks: ie, duration in days / 7; (N, mean, SD, median, and range (minimum, maximum)) will be presented by age group (2-<6 years; 6-<12 years) and overall.

In addition, duration of exposure will be summarized by age group (2-<6 years; 6-<12 years) and overall for the FAS in the following duration categories: <1 week, 1-<2 weeks, 2-<4 weeks, 4-<8 weeks, 8-<12 weeks, 12-<16 weeks, 16-<24 weeks, 24-<32 weeks, 32-<40 weeks and 40-48 weeks.

Total subject years of exposure is calculated as [sum of (days of exposure)/365.25]. Total subject years of exposure will be presented by age group (2-<6 years; 6-<12 years) and overall.

## **4.4.1. Diaries**

A listing will be created for all participants who underwent intensive PK sampling, comprising of the date and time of RPV intake from the start of study treatment (or start of an adjusted RPV-dose, if applicable) until the day of intensive PK sampling, based on the information entered in the participant diary.

#### 4.5. Protocol Deviations

The major protocol deviations may have the potential to impact participants' rights, safety or well-being, or the integrity and/or result of the clinical study. Participants with major protocol deviations will be identified prior to database lock and major protocol deviations (including a category for COVID-19 related protocol deviations) will be summarized by category.

#### 4.6. Prior and Concomitant Medications

Prior medications are defined as any therapy used before the day of first dose (partial or complete) of RPV. Concomitant medications are defined as any therapy used on or after the same day as the first dose of RPV, including those that started before and continue after the first dose of study agent. Follow-up medications are defined as any therapy that started after the date of the last dose of RPV.

For non-ARV therapies, summaries of concomitant medications will be presented by Anatomic and Therapeutic Chemical (ATC) class level using the World Health Organization-Drug Dictionary (WHO-DD), and by age group (2-<6 years; 6-<12 years) and overall. The proportion of participants who receive each concomitant medication will be summarized as well as the proportion of participants who receive at least 1 concomitant medication.

For ARV therapies, summaries of prior and concomitant (ie, background regimen) medications will be presented by individual ARVs and combination ARVs as collected in the electronic Case Report Form (eCRF) by dose and weight group and overall. The proportion of participants for each category of medication will be summarized.

Prior as well as concomitant ARV and concomitant non-ARV therapies will be tabulated. Participants who switched ARV therapy during treatment will be listed.

## 5. EFFICACY

## 5.1. Analysis Specifications

# **5.1.1.** Level of Significance

No statistical testing will be done as this is a single arm trial.

## **5.1.2.** Data Handling Rules

## Viral Load:

Viral load testing will be measured at a central laboratory using standardized HIV-1 viral load assays as the concentration of HIV-1 RNA in plasma. Reanalyzed samples will not be used in any of the calculations or summary statistics.

Imputation of left-censored values: values below the detection limit (ie, 20 copies/ml) will be scored as 1 less than the detection limit in the analysis (ie, 20-1=19 copies/ml), unless explicitly specified differently.

Imputation of right-censored values: in case viral loads were above the upper limit of quantitation, i.e.10,000,000 HIV-1 RNA copies/mL, the viral load will be scored as 1 more than the detection limit in the analysis, unless explicitly specified differently.

If no observation is available at baseline the last available screening value will be taken.

## Immunology:

For cases where <u>no observation is available at the baseline date</u>, the last available screening value will be taken.

In case <u>multiple observations</u> (different sampling dates) are available within a single visit window, only the one closest to the target day will be selected for the displays to select unique observations per time point (visit window).

## **Rounding:**

For point estimates (means or percentages), the following rounding rules are applied:

- CD4 count: 1 decimal
- all other parameters (including viral load in case not log-transformed, and Fold Change (FC)): 1 decimal

For confidence intervals (CIs), median, interquartile range, min and max: number of decimals for according point estimate.

For SDs and SEs: number of decimals for according point estimate + 1 decimal.

## 5.2. Efficacy Endpoints

The following efficacy parameters will be analyzed:

- Virologic outcome (virologic response and virologic failure) applying HIV-1 RNA thresholds 50 and 400 copies/mL using the FDA Snapshot approach, at Week 24/Week 48.
- Change in CD4 cell count (absolute and percentage) from baseline up to Week 24/Week 48.

## **5.2.1.** Definition

Virologic response is defined as follows:

0 = non-responder: the viral load test result is above some threshold value

1 = responder: the viral load test result is below some threshold value

## Virologic failure

**Loss of response:** two consecutive measurements of ≥200 HIV-1 RNA copies/mL at least 2 weeks apart after having been confirmed virologic responder.

Suspected Virologic Failure: HIV-1 RNA ≥200 copies/mL.

# FDA Snapshot approach:

The following outcome subcategories are defined (giving priority in the order as presented below, such that each participant is categorized into a single subcategory)

- 1) Participant's background regimen was switched as not permitted by the protocol; participants who experienced a switch in their background regimen composition that lasted more than one week and not permitted by the protocol (identify these from protocol deviations [ADDV]) and that occurred before the earliest onset of AEs leading to permanent stop, and, if the participant is ongoing, that occurred up to and including the end day of the 24/48 week window, are assigned outcome subcategory = 'Virologic failure switch in background regimen not permitted by the protocol'.
- 2) Participant discontinued trial for virologic failure during treatment phase if reason for discontinuation is 'SUBJECT REACHED A VIROLOGIC ENDPOINT' and HIV-1 RNA is missing at Week 24/48 then outcome subcategory = 'Virologic failure leading to discontinuation';
- 3) Viral load data in the Week 24/48 window
  - if last available HIV RNA in the time window is <50/400 copies/mL then outcome='Virologic success: HIV RNA < 50/400 copies/mL at Week 24/48';
  - if last available HIV RNA in the time window is ≥50/400 copies/mL then outcome='Virologic failure: HIV RNA ≥50/400 copies/mL at Week 24/48;
- 4) No HIV RNA data in Week 24/48 window;
  - if the participant completed Week 24/48 but HIV RNA data at Week 24/48 is missing then outcome='Missing data during window but on study';
  - if the reason for discontinuation='ADVERSE EVENT/HIV RELATED EVENT' and the earliest AE leading to permanent stop was not preceded by a switch in the background regimen that was not permitted by the protocol (see point 1) above), then outcome='Discontinued due to AE/death';
  - if the reason for discontinuation is 'OTHER', 'SPONSORS DECISION', 'SUBJECT DID NOT FULFILL ALL INCLUSION/EXCLUSION CRITERIA', 'SUBJECT INELIGIBLE TO CONTINUE THE TRIAL', 'SUBJECT LOST TO FOLLOW-UP', 'SUBJECT NONCOMPLIANT' or 'SUBJECT WITHDREW CONSENT': if the last available HIV RNA is <50/400 copies/mL (or no post baseline HIV RNA data available), outcome subcategory = 'Discontinued due to other reason and the last available HIV RNA < 50/400 copies/mL, outcome subcategory = 'Virologic failure discontinued due to other reason and last available HIV RNA ≥50/400 copies/mL';

Week 24: The snapshot analysis is based on the last observed viral load data within the Week 24 window (day 141 up to and including day 196, Window 20-28 weeks, baseline = day 1).

Week 48: The snapshot analysis is based on the last observed viral load data within the Week 48 window (day 309 up to and including day 378, Window 44-54 weeks, baseline = day 1).

## **Changes from baseline in CD4+ count:**

The change from baseline in CD4+ count and CD4% at a given time point is defined as: (CD4+/CD4% at a given time point - baseline CD4+/CD4%).

Participants who discontinued will have their CD4+ values after discontinuation imputed with their baseline value, thus resulting in a 0 change; For timepoints with intermittently missing data, last observation carried forward approach is applied (Non-Completer=Failure imputation). Analysis results based on observed data only will also be presented.

For cases where <u>no observation is available at the baseline date</u>, the last available screening value will be taken.

In case <u>multiple observations</u> (different sampling dates) are available within a single visit window, only the one closest to the target day will be selected for the displays to select unique observations per time point (visit window).

The table shell for snapshot analysis will be presented in the DPS.

## 5.2.2. Analysis Methods

Tabulations (numbers and proportions) per time point by age group (2-<6 years; 6-<12 years) and overall for the categorical parameters (virologic response, virologic failures); 95% CIs (Clopper-Pearson) for the virologic response rates over time will be calculated.

Descriptive statistics (n, mean (se), median, and range (minimum and maximum) per time point and graphical display for the continuous parameters CD4<sup>+</sup> cell count and CD4<sup>+</sup> (%) (change from baseline) will be presented. Both observed value as well as imputed values using the NC=F imputation method will be displayed.

Patient profiles will be provided for viral load and CD4+ counts over time.

## 5.3. Other Efficacy Variables

#### 5.3.1. Resistance

## **HIV-1 Viral Genotyping:**

Inclusion of participants for resistance analysis will solely be based on the availability of post-baseline genotypic data within the treatment phase.

The first and the last post-baseline time point within the treatment phase for which genotypic data are available will be analyzed and presented.

Sequencing of HIV-1 protease, reverse transcriptase and integrase will be performed in real time on plasma for participants with (suspected) virologic failure.

## Reverse Transcriptase (RT) resistance associated mutations

- IAS-USA NRTI RAMs (n=22)<sup>2</sup> M41L, A62V, K65E/N/R, D67N, 69ins, K70E/R, L74V, V75I, F77L, Y115F, F116Y, Q151M, M184I/V, L210W, T215F/Y, K219E/Q.
- Extended NNRTI RAMs (n=53)<sup>2</sup> V90I, A98G, L100I, K101E/H/P/Q, K103H/N/S/T, V106A/I/M/T, V108I, E138A/G/K/Q/R, V179D/E/F/G/I/L/T, Y181C/I/V, Y188C/H/L, V189I, G190A/C/E/Q/S/T, H221Y, P225H, F227C/L/R, M230I/L, P236L, K238N/T, L243I, Y318F
- RPV RAMs (n=16) K101E, K101P, E138A, E138G, E138K, E138R, E138Q, V179L, Y181C, Y181I, Y181V, Y188L, H221Y, F227C, M230I, M230L

## Protease resistance associated mutations

- IAS-USA primary PI RAMs (n=24)<sup>2</sup> D30N, V32I, M46I/L, I47A/V, G48V, I50L/V, I54L/M/V, Q58E, T74P, L76V, V82A/F/L/S/T, N83D, I84V, N88S, L90M
- IAS-USA PI RAMs (n = 75)  $^2$  L10C/F/I/R/V, V11I, G16E, K20I/M/R/T/V, L24I, D30N, V32I, L33I/F/V, E34Q, M36I/L/V, K43T, M46I/L, I47A/V, G48V, I50L/V, F53L/Y, I54A/L/M/S/T/V, Q58E, D60E, I62V, L63P, I64L/M/V, H69K/R, A71I/L/T/V, G73A/C/S/T, T74P, L76V, V77I, V82A/F/I/L/S/T, N83D, I84V, I85V, N88D/S, L89I/M/V, L90M, I93L/M

#### Integrase resistance associated mutations (n=27):

- T66A/I/K, L74M, E92G/Q, T97A, G118R, F121Y, E138A/K/T, G140A/C/R/S, Y143C/H/R, S147G, Q148H/K/R, S153F/Y, N155H, R263K

Concordance/discordance with "Virologic Failure" as per FDA Snapshot approach (see section 5.2.1) will be assessed.

Results will be shown in different columns, unless explicitly specified differently in the DPS:

- Non-VF: responder
- Non-VF: discontinued due to AE or other reason
- VF
- Overall

Results from viral genotyping in plasma will be tabulated and described, particularly for participants with virologic failure.

Individual mutations identified via viral genotyping will be reported relative to the HIV-1 WT reference sequence.

## **Retrospective evaluation of RAMs in PBMCs:**

Peripheral Blood Mononuclear Cell (PBMC) sample will be taken to allow retrospective characterization of archived viral resistance, if needed. Inclusion of participants for archived resistance analysis is based on the availability of results obtained at screening, Week 24 or Week 48.

Results from archival viral resistance from PBMC sample will be tabulated and described, particularly for participants with virologic failure.

#### 6. SAFETY

All safety analyses will be based on the FAS. Selected outputs will be generated separately for the first 4 weeks of treatment.

For all continuous safety variables, descriptive statistics will include the N, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized using frequency counts and percentages. For laboratory, ECG and vital sign results, an abnormality is considered treatment-emergent if it is worse than baseline. If baseline is missing, the abnormality is always considered treatment-emergent. For pulse, a shift from 'abnormally low'at baseline to 'abnormally high' post-baseline (or vice versa) is also treatment-emergent.

Safety data will be presented by age group (2-<6 years; 6-<12 years) and overall, unless explicitly specified differently in the DPS.

## 6.1. Adverse Events (AE)

Adverse Event (AE): An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product

The verbatim terms used in the Case Report Form (CRF) by investigators to identify adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA 24.1 or latest).

Any AE occurring at or after the initial administration of RPV through the day of last dose is considered to be treatment emergent. If the event occurs on the day of the initial administration of RPV, and either event time or time of administration are missing, then the event will be assumed to be treatment emergent. If the event date is recorded as partial or completely missing, then the event will be considered to be treatment emergent unless it is known to be prior to the first administration of RPV based on partial onset date or resolution date.

All reported treatment-emergent adverse events will be included in the analysis. For each adverse event, the number and percentage of participants who experience at least 1 occurrence of the given event will be summarized by age group (2-<6 years; 6-<12 years) and overall.

Summary tables will be provided for all treatment-emergent:

- AEs
- SAEs
- AEs leading to discontinuation of RPV
- AEs leading to dose interruption of RPV
- AEs by severity
- AEs by relationship to RPV

In addition to the summary tables, listings will be provided for participants who had:

- SAEs
- AEs leading to discontinuation of RPV

- HIV-related AEs
- Stage 3-defining Opportunistic Illnesses in HIV infection (see Attachment 3: STAGE-3-DEFINING OPPORTUNISTIC ILLNESSES IN HIV INFECTION)

A listing of participants who died during the study will be provided.

Overall AE summary tables by preferred term/SOC for SAEs and pregnancies, AEs leading to discontinuation, AEs at least grade 3, HIV-related AEs, stage 3-defining Opportunistic Illnesses in HIV infection and AEs at least possibly related to RPV will be presented throughout the treatment phase only; any AEs in the Follow-up phase will be listed only.

## Number of occurrences of an AE:

Number of recorded events of the same preferred term, during the trial phase. Combined events (i.e. within the same phase) will be counted only once.

## AE grading:

Reported AEs parameters and grades are based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (ATTACHMENT 1: DAIDS GRADING TABLE).

#### AE duration.

For the calculation of duration of AEs, only AEs are considered with complete start and end date or for which the end date is imputed (see STEP 1 for imputation of end date). Duration is calculated as End date – Start date +1

## Onset day of AE:

- *after start of investigational medication* = first start date of the AE first intake date of investigational medication + 1 day. In case of combined events, the onset day will be computed only once, and relative to the start date of the first event.
- *in the phase* = first start date of the AE start date of the phase in which the AE emerges + 1 day. In case of combined events, the onset day will be computed only once, and relative to the start date of the first event.

## Adverse Events of Interest (EOI):

Different events of interest will be investigated separately. A list of Events of Interest (EOI) is maintained at Janssen Infectious Diseases which is updated (if necessary) based on accumulating AE data from both RPV Adult Phase III studies. A list of EOI for analysis purposes will be provided prior to the database lock. The different classes of events of interest that should be investigated are the following:

- <u>Skin events of interest:</u> The skin events of interest will be defined based on the adverse event preferred terms and will be summarized using alternative groupings: 'Dermatitis Contact', 'Dermatitis / Eczema', 'Oedema', 'Rash', 'Rash Vesicular', 'Other'.
- Neuropsychiatric events of interest: Neuropsychiatric events of interest will be defined based on
  the adverse event preferred terms and will be summarized using alternative groupings: 'Nervous
  System Disorders', 'Psychiatric Disorders'. Under the 'Psychiatric Disorders' an extra row will
  be included, namely the combination of "ABNORMAL DREAMS" or "NIGHTMARES".
- <u>Potential QT prolongation-related events:</u> selection of preferred terms is based on a MedDRA standardized query for "Torsade de pointes/OT prolongation"
- <u>Hepatic events of interest:</u> Hepatic events of interest will be defined based on the adverse event preferred terms.

- Endocrinology events of interest: These are defined as all endocrinology events categorized under the system organ class 'ENDOCRINE DISORDERS' or all AEs categorized under the system organ class 'INVESTIGATIONS' related to any of the endocrine analytes measures (cortisol, 17-OH progesterone, aldosterone, dehydroepiandrosterone (DHEAS), androstenedione, testosterone) in the trial.
- <u>AIDS defining Illnesses and Stage-3-defining Opportunistic Illnesses in HIV Infection:</u> All adverse events classified as CDC Stage 3 and Stage-3-defining Opportunistic Illnesses.

## **6.2.** Clinical Laboratory Tests

All clinical laboratory tests will be displayed for the participants included in the FAS. Results from central laboratory testing (Covance/Labcorp) will be included in the analysis; results from local laboratories will not be included in the analysis, only listed.

Observed and change from baseline to each scheduled time point will be summarized descriptively for laboratory tests and displayed by age group (2-<6 years; 6-<12 years) and overall.

The laboratory tests will be grouped as follows:

- 1) General biochemistry (albumin, blood urea nitrogen, calcium, calcium adjusted for albumin, chloride, phosphate, creatinine, potassium, sodium, uric acid, creatinine phosphokinase, ...)
- 2) Pancreatic Parameters (pancreatic amylase, lipase)
- 3) Renal Parameters (serum creatinine, eGFR (creatinine), ...)
- 4) Hepatic parameters (ALT, AST, gamma-GT, alkaline phosphatase, LDH, bilirubin (all types), total protein...)
- 5) Lipids and glucose (cholesterol, HDL cholesterol (HDL-C) (all types), LDL cholesterol (LDL-C) (all types), TC/HDL-C, insulin, glucose, triglycerides, ...)
- 6) General hematology (Hematocrit, hemoglobin, red blood cell count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH) and mean corpuscular hemoglobin concentration (MCHC), platelet count, white blood cell count)
- 7) Hematology differential counts (Basophils, eosinophils, lymphocytes, monocytes, neutrophils (counts and %), ...)
- 8) Endocrinology (Cortisol, 17-hydroxyprogesterone, dehydroepiandrosterone (DHEAS), androstenedione, testosterone, follicle stimulating hormone (FSH), luteinizing hormone (LH))

#### **Toxicity grades:**

Toxicity grades are determined according to the <u>DAIDS grading list</u> (ATTACHMENT 1: DAIDS GRADING TABLE). In case no toxicity grades are defined for a test, the abnormalities (above/below normal range) are used. In determining toxicity grades, the following rules are applied:

- Laboratory values are <u>rounded</u> to the same number of decimals as the DAIDS grading, and the rounded value is used to allocate a grading to the value.
- There is no overruling of the DAIDS grades when the value is between the normal limits
- In case no numeric value is available, but only a verbatim term (e.g. PTT>120) then the numeric value will be derived by determining the closest value to the cut-off value, taking into account the usual number of decimals for the particular parameter, in order to be able to allocate a grade to these observations.

Note: as the grading scale for some parameters in the DAIDS grading table has some gaps (zones where no toxicity grade definition exists), laboratory results falling in these zones are allocated to the immediate worst-case grade.

Cross-tabulations for the worst toxicity grades versus reference per laboratory test will be reported.

## Endocrine safety: Adrenocorticotropic hormone (ACTH) stimulation testing

## Abnormal ACTH response:

The ACTH test result will be categorized into the following categories:

- 1) Maximum cortisol measurement (time points T0 and T60) ≥ 500 nmol/L
- 2) Maximum cortisol measurement (time points T0 and T60) [450; 500[ nmol/L
- 3) Maximum cortisol measurement (time points T0 and T60) < 450 nmol/L

Cross-tabulations for on-treatment ACTH stimulation test abnormalities (defined as cortisol after ACTH stimulation < 500 nmol/L) will be reported for following time points: last on-treatment measurement, worst on-treatment measurement.

Endocrine safety (cortisol and 17-hydroxyprogesterone) will be summarized per analysis time point for following measurements: T0, T60. In addition, abnormal basal cortisol (defined as <248 nmol/L) will be tabulated per analysis time point.

## 6.3. Vital Signs and Physical Examination Findings

Continuous vital sign parameters including height, weight, pulse, blood pressure (systolic and diastolic), and BMI will be summarized at each assessment time point. BMI will be calculated as weight (kg)/(height (m))<sup>2</sup>, at each time point that body weight is measured.

Observed and change from baseline will be summarized by age group (2-<6 years; 6-<12 years) and overall. Descriptive statistics (mean, standard deviation, median, minimum and maximum) will be presented.

Incidence of markedly abnormal vital signs while on treatment, as defined in Table 5, will be summarized for participants who had a baseline assessment and at least 1 postbaseline assessment for that vital sign.

**Table 5: Markedly Abnormal Vital Signs** 

| Vital Sign | Criteria |
|---|---|
| Pulse | ≥ 120 bpm for higher limit |
| | ≤ 50 bpm for lower limit |
| Systolic blood pressure | Grade 1: >120 mmHg |
| | Grade 2: ≥95 <sup>th</sup> to <99 <sup>th</sup> percentile +5 mmHg adjusted for age, height, and gender (systolic and/or diastolic) |
| | Grade 3: ≥99th percentile +5 mmHg adjusted for age, height, and gender (systolic and/or diastolic) |
| Diastolic blood pressure | Grade 1: >80 mmHg |
| Grade 2: ≥95 <sup>th</sup> to <99 <sup>th</sup> percentile +5 mmHg adjusted for age, he gender (systolic and/or diastolic) | |
| | Grade 3: ≥99th percentile +5 mmHg adjusted for age, height, and gender (systolic and/or diastolic) |

23

To classify vital sign measurements into abnormality codes, the following approach is used:

An absolute blood pressure measurement is translated into a blood pressure percentile (cf table provided in Attachment 2: BLOOD PRESSURE LEVELS BY AGE AND HEIGHT PERCENTILES) based on the participant's age and height percentile (= height-for-age percentiles at the time of the blood pressure measurement).

For calculation of height-for-age percentiles, see SAS programs available from http://www.who.int/childgrowth/software/en/ (up to 5 years of age) and http://www.who.int/growthref/tools/en/ (from 5 to 19 years of age).

Last-Observation-Carried-Forward (LOCF) imputation will be used for missing height percentiles. In case a participant's height percentile does not exactly match a value reported in attachment 2, calculated height-for-age percentiles are translated into values available in attachment 2 as follows:

| Calculated height-for-age percentile | Height Percentile |
|--------------------------------------|-------------------|
| 1 - 7 | 5 |
| 8 - 17 | 10 |
| 18 - 37 | 25 |
| 38 - 62 | 50 |
| 63 - 82 | 75 |
| 83 - 92 | 90 |
| 93 - 100 | 95 |

Also, occurrence of orthostatic hypotension will be summarized, defined as:

supine SBP – standing SBP  $\geq$  20 mmHg OR supine DBP – standing DBP  $\geq$  10 mmHg

#### **Physical Examination:**

Physical examination findings will be summarized at each scheduled time point with full physical examination per body system by age group (2-<6 and 6-<12 years) and overall.

Physical examination abnormalities will be listed.

## **Growth Examination:**

Growth will be followed regularly and evaluated consistently using WHO standardized growth charts, using age at visit.

- Height (cm)
- Height-for-age (z-score and percentile)
- Weight (kg)
- Weight-for-age (z-score and percentile)
- BMI = weight  $(kg)/(height (m))^2$
- BMI-for-age (z-score and percentile)

Observed and change from baseline will be summarized for by age group (2-<6 and 6-<12 years) and overall. Descriptive statistics (mean, standard deviation, median, minimum and maximum) will be presented.

## **Tanner Stage:**

Tanner stage (for pubic hair and genitalia/breasts) will be cross-tabulated versus baseline by age. In addition, in girls, the occurrence of first menses during treatment will also be cross-tabulated versus baseline, and the date of menarche will be listed.

## 6.4. Electrocardiogram

All ECG parameters will be displayed for the participants included in the FAS. No statistical testing will be performed. In addition, for QTcB/F at pre-dose and post-dose at Week 4, 24, and 48 will be analyzed as separate time points.

The ECG parameters that will be analyzed are heart rate, PR interval, RR interval, QRS interval, QT interval, QTcB and QTcF using the following correction methods: Bazett's formula (QTcB), Fridericia's formula (QTcF).

Bazett's formula: QTcB (ms) = 
$$\frac{QT(ms)}{\sqrt{RR(ms)/1000}}$$

Fridericia's formula: QTcF (ms) = 
$$\frac{QT(ms)}{\sqrt[3]{RR(ms)/1000}}$$

\* If RR is missing, it will be derived from HR (see formula below) if this is parameter is available from the same ECG reading as the QT. HR from the Vital Signs dataset will not be used to calculate the corrected QT parameters.

$$RR(ms)$$
 1000\* $\frac{60}{HR(bpm)}$ 

QT corrections will be re-computed even if they are provided.

Observed and change from baseline to each scheduled time point will be descriptively summarized by dose and weight group and overall for the above ECG parameters.

A listing of clinically relevant ECG results will also be provided.

The number and percentage of participants within each of the categories defined below will be presented for the maximum postbaseline value (ie: the maximum ECG result over the study period) by dose and weight group, and overall.

Categories to assess QT prolongation:

QTc Interval: QTcB criteria are based on DAIDS 2017 (see the study protocol Addendum 2: DAIDS Table) and QTcF criteria are from MOCHA/CRAYON protocol:

• Normal:

QTcF: <460 ms OTcB: <450 ms

• Grade 1:

QTcF:  $\ge$ 460 to  $\le$ 480 ms QTcB:  $\ge$ 450 to  $\le$ 470 ms

• Grade 2:

QTcF:  $\ge$ 480 to < 500 ms QTcB:  $\ge$ 470 to  $\le$  500 ms

#### • Grade 3:

QTcF:  $\geq$ 500 ms OR QTcF  $\geq$ 480 ms AND QTcF > 60 ms greater than baseline QTcB: >500 ms OR QTcB  $\geq$  60 ms greater than baseline

#### • Grade 4:

QTcF/B: Life-threatening consequences: eg, Torsades de pointes, other serious ventricular dysrhythmias.

## QTcF change from baseline:

• normal: <30 ms

• borderline: >30 to <60 ms

• abnormal high: >60 ms

## QTcB change from baseline:

• normal: <30 ms

• borderline:  $\geq$ 30 to  $\leq$ 60 ms

• abnormal high: >60 ms

#### 7. PHARMACOLOGY

## 7.1. Population Pharmacokinetics

Population pharmacokinetic parameters (AUC<sub>24h</sub> and  $C_{0h}$ ; based on sparse sampling) will be available for all participants.

# Pharmacokinetic/Pharmacodynamic Relationships

## PK and Efficacy

Scatterplot of individual PK parameters (AUC<sub>24h</sub> and C<sub>0h</sub>) by virologic response (plasma viral load <50/400 copies/mL) as well as virologic failure (HIV RNA  $\ge$ 50/400 copies/mL) using FDA Snapshot (yes/no) at Week 24/Week 48, will be created.

## PK and Safety

Relationship between RPV pharmacokinetics ( $AUC_{24h}$  only) and the following AE groups / abnormalities will be explored graphically by the means of scatterplots.

- Rash (yes/no) (The skin event of interest alternative grouping of 'Rash' will be used.)
- All neuropsychiatric events of interest combined (yes/no)
- Combined AEs in the Nervous System Disorders alternative grouping (yes/no)
- Combined AEs in the 'Psychiatric Disorders' SOC (yes/no)
- Combined AEs in the 'Gastrointestinal Disorders' SOC (yes/no)
- Combined AEs in the 'Blood and Lymphatic Disorders' SOC (yes/no)
- Combined AEs with preferred terms 'abnormal dreams', 'vivid dreams', 'nightmare' (yes/no)
- Dizziness (yes/no)
- Headache (yes/no)
- QTcF abnormalities (yes/no), both based on absolute values and changes from baseline (section 6.4)

Scatterplots of individual PK parameter values (AUC<sub>24h</sub> only) by specific laboratory/ECG parameters (change from baseline), presented in the following table, will be shown.

| Biochemistry | Lipids | Hematology | Glucose<br>metabolism | ECG |
|---|---|---|---|---|
| ALT ([max]) | HDL ([min]) | Hemoglobin ([min]) | Glucose ([max]) | QTcF<br>([max]) |
| AST ([max]) Total bilirubin ([max]) Alkaline phosphatase ([max]) Pancreatic amylase ([max]) Lipase ([max]) Creatinine ([max]) eGFR (creatinine) ([min]) | LDL ([max]) Triglycerides ([max]) Total cholesterol ([max]) Total cholesterol / HDL ([min]) | Hematocrit ([min]) | Insulin ([min])<br>HOMA-IR ([max]) | (L J) |

| Endocrine (Cortisol, 17-OH Progesterone) | | |
|---|---|---|
| Cortisol | 17-OH Progesterone | Aldosterone |
| morning/T0 (non-ACTH) | morning/T0 (non-ACTH) | morning/T0 (non-ACTH) ([min]) |
| ([min]) | ([max]) | |

[min] or [max] indicates which value to use, i.e. either the smallest or largest value respectively

## 7.2. Other Pharmacology Endpoints

## Palatability:

The palatability of the 2.5 mg RPV tablet formulation will be assessed in a palatability questionnaire after a 2-week treatment period by documenting the participant's perception using a 5-point hedonic scale.

The number and percentage of participants within each of the categories, as well as cumulatively (from best to worst) will be presented by age group (2-<6 years; 6-<12 years) and overall.

## **Swallowability:**

The swallowability of the RPV 25-mg tablet formulation will be assessed in a swallowability questionnaire after a 2-week treatment period by documenting the participant's reaction when he or she is given the 25 mg tablet formulation of RPV medication.

The number and percentage of participants within each of the response to two questions (ease of swallowing, acceptability longer term) will be presented by age group (2-<6 years; 6-<12 years) and overall.

Similarly, responses by the observer (how tablet was taken, reported problems, whether second attempt was needed) will be tabulated.

## **REFERENCES**

- 1. http://www.cdc.gov/growthcharts
- 2. Wensing AM, Calvez V, Ceccherine-Silberstein, et al. 2019 update of the drug resistance mutations in HIV-1. Top Antivir Med Sep/Oct 2019; 27(3):111-121
- 3. NPR-20060022-VRR v7.0
- 4. Bennett DE, Camacho RJ, Otelea D, Kuritzkes DR, Fleury H, et al. 2009 Drug Resistance Mutations for Surveillance of Transmitted HIV-1 Drug-Resistance: 2009 Update. PLoS ONE 4(3): e4724. doi:10.1371/journal.pone.000472
- 5. H C Bazett: An analysis of the time-relations of electrocardiogram; Heart 1920; 7: 353 370.
- 6. L S Fridericia: Die systolendauer im elektrokardiogramm bei normalen menchen und bei herzkranken; Acta Med Scand 1920; 15: 335 642.

Approved, Date: 27 March 2023

## **ATTACHMENTS**

## ATTACHMENT 1: DAIDS GRADING TABLE

DIVISION OF AIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS, CORRECTED VERSION 2.1, PUBLISH DATE: JULY 2017

| | LABORATORY VALUES <sup>III</sup> | | | |
|---|---|---|---|---|
| | | CHEMISTRIES | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Acidosis | NA | pH ≥7.3 to <lln< td=""><td>pH &lt;7.3 without<br/>life-threatening<br/>consequences</td><td>pH &lt;7.3 with<br/>life-threatening<br/>consequences</td></lln<> | pH <7.3 without<br>life-threatening<br>consequences | pH <7.3 with<br>life-threatening<br>consequences |
| Albumin, Low (g/dL; g/L) | 3.0 to <lln<br>30 to <lln< td=""><td>≥2.0 to &lt;3.0<br/>≥20 to &lt;30</td><td>&lt;2.0<br/>&lt;20</td><td>NA</td></lln<></lln<br> | ≥2.0 to <3.0<br>≥20 to <30 | <2.0<br><20 | NA |
| ALP, High | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Alkalosis | NA | pH >ULN to ≤7.5 | pH >7.5 without<br>life-threatening<br>consequences | pH >7.5 with<br>life-threatening<br>consequences |
| ALT or SGPT, High<br>Report only 1 | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Amylase (Pancreatic)<br>or Amylase (Total),<br>High<br>Report only 1 | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| AST or SGOT, High<br>Report only 1 | 1.25 to <2.5×ULN | 2.5 to <5.0×ULN | 5.0 to <10.0×ULN | ≥10.0×ULN |
| Bicarbonate, Low<br>(mEq/L; mmol/L) | 16.0 to <lln<br>16.0 to <lln< td=""><td>11.0 to &lt;16.0<br/>11.0 to &lt;16.0</td><td>8.0 to &lt;11.0<br/>8.0 to &lt;11.0</td><td>&lt;8.0<br/>&lt;8.0</td></lln<></lln<br> | 11.0 to <16.0<br>11.0 to <16.0 | 8.0 to <11.0<br>8.0 to <11.0 | <8.0<br><8.0 |
| Bilirubin<br>Direct Bilirubin <sup>n</sup> ,<br>High<br>aged >28 days | NA | NA | >ULN with other signs<br>and symptoms of<br>hepatotoxicity | >ULN with<br>life-threatening<br>consequences<br>(eg, signs and<br>symptoms of liver<br>failure) |
| aged ≤28 days | ULN to ≤1 mg/dL | >1 to ≤1.5 mg/dL | >1.5 to ≤2 mg/dL | >2 mg/dL |
| Total Bilirubin, High<br>aged >28 days | 1.1 to <1.6×ULN | 1.6 to <2.6×ULN | 2.6 to <5.0×ULN | ≥5.0×ULN |
| aged ≤28 days | NA | NA | NA | NA |

mEq=milliequivalent, LLN=lower limit of normal, NA=not applicable, SGOT=serum glutamic-oxaloacetic transaminase, SGPT=serum glutamate-pyruvate transaminase

m Reminder: An asymptomatic abnormal laboratory finding without an accompanying AE should not be reported to DAIDS in an expedited time frame unless it meets protocol-specific reporting requirements.

n Direct bilirubin >1.5 mg/dL in a participant aged <28 days should be graded as grade 2, if <10% of the total bilirubin.

## Statistical Analysis Plan TMC278HTX2002 (W24 &W48 Analysis)

| Calcium, High | | | | |
|---|---|---|---|---|
| (mg/dL; mmol/L) | 10.6 to <11.5 | 11.5 to <12.5 | 12.5 to <13.5 | ≥13.5 |
| aged ≥7 days | 2.65 to <2.88 | 2.88 to <3.13 | 3.13 to <3.38 | ≥3.38 |
| aged <7 days | 11.5 to <12.4 | 12.4 to <12.9 | 12.9 to <13.5 | ≥13.5 |
| ugeu uuys</td <td>2.88 to &lt;3.10</td> <td>3.10 to &lt;3.23</td> <td>3.23 to &lt;3.38</td> <td>≥3.38</td> | 2.88 to <3.10 | 3.10 to <3.23 | 3.23 to <3.38 | ≥3.38 |
| 61: 6: 8 | | | | |
| Calcium (Ionized), | >ULN to <6.0 | 6.0 to <6.4 | 6.4 to <7.2 | ≥7.2 |
| High | >ULN to <1.5 | 1.5 to <1.6 | 1.6 to <1.8 | ≥1.8 |
| (mg/dL; mmol/L) | | | | |
| Calcium, Low | | | | |
| (mg/dL; mmol/L) | 7.8 to < 8.4 | 7.0 to <7.8 | 6.1 to < 7.0 | <6.1 |
| aged ≥7 days | 1.95 to <2.10 | 1.75 to <1.95 | 1.53 to <1.75 | < 1.53 |
| aged <7 days | 6.5 to <7.5 | 6.0 to <6.5 | 5.50 to <6.0 | <5.50 |
| agea adys</td <td>1</td> <td>1</td> <td></td> <td>&lt;1.38</td> | 1 | 1 | | <1.38 |
| | 1.63 to <1.88 | 1.50 to <1.63 | 1.38 to <1.50 | |
| Calcium (Ionized), | <lln 4.0<="" td="" to=""><td>3.6 to &lt;4.0</td><td>3.2 to &lt;3.6</td><td>&lt;3.2</td></lln> | 3.6 to <4.0 | 3.2 to <3.6 | <3.2 |
| Low | <lln 1.0<="" td="" to=""><td>0.9 to &lt;1.0</td><td>0.8 to &lt; 0.9</td><td>&lt; 0.8</td></lln> | 0.9 to <1.0 | 0.8 to < 0.9 | < 0.8 |
| (mg/dL; mmol/L) | | | | |
| Cardiac Troponin I, | NA | NA | NA | Levels consistent with |
| High | | | | myocardial infarction |
| | | | | or unstable angina as |
| | | | | defined by the local |
| | | | | laboratory |
| C T2 | 2. 6.7737 | 6. 40.7737 | 10. 00. 7777 | _ |
| Creatine Kinase, | 3 to <6×ULN | 6 to <10×ULN | 10 to <20×ULN | ≥20×ULN |
| High | | | | |
| Creatinine, High | 1.1 to 1.3×ULN | >1.3 to 1.8×ULN OR | >1.8 to <3.5×ULN OR | ≥3.5×ULN OR |
| Report only 1° | | Increase to 1.3 to | Increase to 1.5 to | Increase of |
| | | <1.5×participant's | <2.0×participant's | ≥2.0×participant's |
| | | baseline | baseline | baseline |
| Creatinine | NA | <90 to 60 ml/min or | <60 to 30 ml/min or | <30 ml/min or |
| Clearance <sup>p</sup> or eGFR, | | ml/min/1.73 m <sup>2</sup> OR | ml/min/1.73 m <sup>2</sup> OR | ml/min/1.73 m <sup>2</sup> OR |
| Low | | 10% to <30% decrease | 30% to <50% decrease | ≥50% decrease from |
| Report only 1° | | from participant's | from participant's | participant's baseline |
| Report only 1 | | baseline | baseline | or dialysis needed |
| | | Oascillic | Oascillic | or marysis ficeucu |
| Glucose | | | | |
| (mg/dL; mmol/L) | | | | |
| Fasting, High | 110 to 125 | >125 to 250 | >250 to 500 | ≥500 |
| | 6.11 to < 6.95 | 6.95 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Nonfasting, High | 116 to 160 | >160 to 250 | >250 to 500 | ≥500 |
| | 6.44 to <8.89 | 8.89 to <13.89 | 13.89 to <27.75 | ≥27.75 |
| Glucose, Low | | | | |
| (mg/dL; mmol/L) | 55 to 64 | 40 to <55 | 30 to <40 | <30 |
| aged ≥1 month | 3.05 to <3.55 | 2.22 to <3.05 | 1.67 to <2.22 | <1.67 |
| aged <1 month | 50 to 54 | 40 to <50 | 30 to <40 | <30 |
| agea <1 month | | | | |
| | 2.78 to <3.00 | 2.22 to <2.78 | 1.67 to <2.22 | <1.67 |
| Lactate, High | ULN to <2.0×ULN | ≥2.0×ULN without | Increased lactate with | Increased lactate with |
| | without acidosis | acidosis | pH <7.3 without | pH <7.3 with |
| | | | life-threatening | life-threatening |
| | | | consequences | consequences |

LLN=lower limit of normal, NA=not applicable

o Reminder: Choose the method that selects for the higher grade.

Use the applicable formula (ie, Cockroft-Gault in mL/min or Schwartz, modification of diet in renal disease study [MDRD], or chronic kidney disease epidemiology collaboration [CKD-Epi] in mL/min/1.73m²). Sites should choose the method defined in their study and when not specified, use the method most relevant to the study population.

| | LABORATORY VALUES | | | |
|---|---|---|---|---|
| | | CHEMISTRIES | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Lipase, High | 1.1 to <1.5×ULN | 1.5 to <3.0×ULN | 3.0 to <5.0×ULN | ≥5.0×ULN |
| Lipid Disorders<br>(mg/dL; mmol/L)<br>Cholesterol, Fasting,<br>High<br>aged ≥18 years | 200 to <240<br>5.18 to <6.19 | 240 to <300<br>6.19 to <7.77 | ≥300<br>≥7.77 | NA |
| aged <18 years | 170 to <200<br>4.40 to <5.15 | 200 to <300<br>5.15 to <7.77 | ≥300<br>≥7.77 | NA |
| LDL, Fasting, High | 130 to <160 | 160 to <190 | ≥190 | NA |
| aged ≥18 years | 3.37 to <4.12 | 4.12 to <4.90 | ≥4.90 | |
| aged >2 to | 110 to <130 | 130 to <190 | ≥190 | NA |
| <18 years | 2.85 to <3.34 | 3.34 to <4.90 | ≥4.90 | |
| Triglycerides, | 150 to 300 | >300 to 500 | >500 to <1,000 | >1,000 |
| Fasting, High | 1.71 to 3.42 | >3.42 to 5.7 | >5.7 to 11.4 | >11.4 |
| Magnesium <sup>q</sup> , Low | 1.2 to <1.4 | 0.9 to <1.2 | 0.6 to <0.9 | <0.6 |
| (mEq/L; mmol/L) | 0.60 to <0.70 | 0.45 to <0.60 | 0.30 to <0.45 | <0.30 |
| Phosphate, Low<br>(mg/dL; mmol/L)<br>aged >14 years | 2.0 to <lln<br>0.65 to <lln< td=""><td>1.4 to &lt;2.0<br/>0.45 to &lt;0.65</td><td>1.0 to &lt;1.4<br/>0.32 to &lt;0.45</td><td>&lt;1.0<br/>&lt;0.32</td></lln<></lln<br> | 1.4 to <2.0<br>0.45 to <0.65 | 1.0 to <1.4<br>0.32 to <0.45 | <1.0<br><0.32 |
| aged 1 to | 3.0 to <3.5 | 2.5 to <3.0 | 1.5 to <2.5 | <1.5 |
| 14 years | 0.97 to <1.13 | 0.81 to <0.97 | 0.48 to <0.81 | <0.48 |
| aged <1 year | 3.5 to <4.5 | 2.5 to <3.5 | 1.5 to <2.5 | <1.5 |
| | 1.13 to <1.45 | 0.81 to <1.13 | 0.48 to <0.81 | <0.48 |
| Potassium, High | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| (mEq/L; mmol/L) | 5.6 to <6.0 | 6.0 to <6.5 | 6.5 to <7.0 | ≥7.0 |
| Potassium, Low | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| (mEq/L; mmol/L) | 3.0 to <3.4 | 2.5 to <3.0 | 2.0 to <2.5 | <2.0 |
| Sodium, High | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| (mEq/L; mmol/L) | 146 to <150 | 150 to <154 | 154 to <160 | ≥160 |
| Sodium, Low | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| (mEq/L; mmol/L) | 130 to <135 | 125 to <130 | 121 to <125 | ≤120 |
| Uric Acid, High | 7.5 to <10.0 | 10.0 to <12.0 | 12.0 to <15.0 | ≥15.0 |
| (mg/dL; mmol/L) | 0.45 to <0.59 | 0.59 to <0.71 | 0.71 to <0.89 | ≥0.89 |

LDL=low-density lipoprotein, LLN=lower limit of normal, mEq=milliequivalent, NA=not applicable q To convert a magnesium value from mg/dL to mmol/L, laboratories should multiply by 0.4114.

| Absolute CD4 <sup>+</sup><br>Count, Low<br>(cells/mm <sup>3</sup> ; cells/L) | 300 to <400 | 200 to <300 | 100 to <200 | <100 |
|---|---|---|---|---|
| aged > 5 years (not<br>HIV-infected) | 0.300×10° to<br><0.400×10° | 0.200×10° to<br><0.300×10° | 0.100×10° to<br><0.200×10° | <0.100×10° |
| Absolute Lymphocyte<br>Count, Low | | | | |
| (cells/mm³; cells/L)<br>aged >5 years<br>(not HIV-infected) | 600 to <650<br>0.600×10 <sup>9</sup> to<br><0.650×10 <sup>9</sup> | 500 to <600<br>0.500×10° to<br><0.600×10° | 350 to <500<br>0.350×10 <sup>9</sup> to<br><0.500×10 <sup>9</sup> | <350<br><0.350×10° |
| Absolute Neutrophil | | | | |
| Count, Low<br>(cells/mm³; cells/L)<br>aged >7 days | 800 to 1,000<br>0.800×10 <sup>9</sup> to<br>1.000×10 <sup>9</sup> | 600 to 799<br>0.600×10 <sup>9</sup> to<br>0.799×10 <sup>9</sup> | 400 to 599<br>0.400×10 <sup>9</sup> to<br>0.599×10 <sup>9</sup> | <400<br><0.400×10° |
| aged 2 to 7 days | 1,250 to 1,500<br>1.250×10 <sup>9</sup> to<br>1.500×10 <sup>9</sup> | 1,000 to 1,249<br>1.000×10 <sup>9</sup> to<br>1.249×10 <sup>9</sup> | 750 to 999<br>0.750×10 <sup>9</sup> to<br>0.999×10 <sup>9</sup> | <750<br><0.750×10° |
| aged ≤1 day | 4,000 to 5,000<br>4.000×10 <sup>9</sup> to<br>5.000×10 <sup>9</sup> | 3,000 to 3,999<br>3.000×10 <sup>9</sup> to<br>3.999×10 <sup>9</sup> | 1,500 to 2,999<br>1.500×10 <sup>9</sup> to<br>2.999×10 <sup>9</sup> | <1,500<br><1.500×10° |
| Fibrinogen,<br>Decreased<br>(mg/dL; g/L) | 100 to <200<br>1.00 to <2.00<br>OR<br>0.75 to <1.00×LLN | 75 to <100<br>0.75 to <1.00<br>OR<br>≥0.50 to <0.75×LLN | 50 to <75<br>0.50 to <0.75<br>OR<br>0.25 to <0.50×LLN | <50<br><0.50<br>OR<br><0.25×LLN<br>OR Associated with<br>gross bleeding |
| Hemoglobin <sup>r</sup> , Low | | | | |
| (g/dL; mmol/L) <sup>s</sup><br>aged ≥13 years<br>(male only) | 10.0 to 10.9<br>6.19 to 6.76 | 9.0 to <10.0<br>5.57 to <6.19 | 7.0 to <9.0<br>4.34 to <5.57 | <7.0<br><4.34 |
| aged ≥13 years<br>(female only) | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| aged 57 days to<br><13 years (male<br>and female) | 9.5 to 10.4<br>5.88 to 6.48 | 8.5 to <9.5<br>5.25 to <5.88 | 6.5 to <8.5<br>4.03 to <5.25 | <6.5<br><4.03 |
| aged 36 to 56 days<br>(male and female) | 8.5 to 9.6<br>5.26 to 5.99 | 7.0 to <8.5<br>4.32 to <5.26 | 6.0 to <7.0<br>3.72 to <4.32 | <6.0<br><3.72 |
| aged 22 to 35 days<br>(male and female) | 9.5 to 11.0<br>5.88 to 6.86 | 8.0 to <9.5<br>4.94 to <5.88 | 6.7 to <8.0<br>4.15 to <4.94 | <6.7<br><4.15 |
| aged 8 to ≤21 days<br>(male and female) | 11.0 to 13.0<br>6.81 to 8.10 | 9.0 to <11.0<br>5.57 to <6.81 | 8.0 to <9.0<br>4.96 to <5.57 | <8.0<br><4.96 |
| aged ≤7 days (male<br>and female) | 13.0 to 14.0<br>8.05 to 8.72 | 10.0 to <13.0<br>6.19 to <8.05 | 9.0 to <10.0<br>5.59 to <6.19 | <9.0<br><5.59 |

#### LLN=lower limit of normal

r Male and female sex are defined as sex at birth. For transgender participants aged ≥13 years who have been on hormone therapy for more than 6 consecutive months, grade hemoglobin based on the gender with which they identify (ie, a transgender female should be graded using the female sex at birth hemoglobin laboratory values).

s The most commonly used conversion factor to convert g/dL to mmol/L is 0.6206. For grading hemoglobin results obtained by an analytic method with a conversion factor other than 0.6206, the result must be converted to g/dL using the appropriate conversion factor for the particular laboratory.

| | | LABORATORY VALU | ES | |
|---|---|---|---|---|
| HEMATOLOGY | | | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| INR, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.5×ULN | 1.5 to <2.0×ULN | 2.0 to <3.0×ULN | ≥3.0×ULN |
| Methemoglobin<br>(% hemoglobin) | 5.0% to <10.0% | 10.0% to <15.0% | 15.0% to <20.0% | ≥20.0% |
| PTT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.66×ULN | 1.66 to <2.33×ULN | 2.33 to <3.00×ULN | ≥3.00×ULN |
| Platelets, Decreased (cells/mm³; cells/L) | 100,000 to <125,000<br>100.000×10 <sup>9</sup> to<br><125.000×10 <sup>9</sup> | 50,000 to <100,000<br>50.000×10° to<br><100.000×10° | 25,000 to <50,000<br>25.000×10° to<br><50.000×10° | <25,000<br><25.000×10° |
| PT, High<br>(not on anticoagulation<br>therapy) | 1.1 to <1.25×ULN | 1.25 to <1.50×ULN | 1.50 to <3.00×ULN | ≥3.00×ULN |
| WBC, Decreased<br>(cells/mm³; cells/L)<br>aged >7 days | 2,000 to 2,499<br>2.000×10 <sup>9</sup> to<br>2.499×10 <sup>9</sup> | 1,500 to 1,999<br>1.500×10 <sup>9</sup> to<br>1.999×10 <sup>9</sup> | 1,000 to 1,499<br>1.000×10 <sup>9</sup> to<br>1.499×10 <sup>9</sup> | <1,000<br><1.000×10° |
| aged ≤7 days | 5,500 to 6,999<br>5.500×10° to<br>6.999×10° | 4,000 to 5,499<br>4.000×10° to<br>5.499×10° | 2,500 to 3,999<br>2.500×10 <sup>9</sup> to<br>3.999×10 <sup>9</sup> | <2,500<br><2.500×10° |

INR=International Normalized Ratio, NA=not applicable, PT=prothrombin time, PTT=partial thromboplastin time

| | LABORATORY VALUES | | | |
|---|---|---|---|---|
| | URINALYSIS | | | |
| PARAMETER | GRADE 1<br>MILD | GRADE 2<br>MODERATE | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
| Glycosuria<br>(random collection<br>tested by dipstick) | Trace to 1+ or<br>≤250 mg | 2+ or >250 to ≤500 mg | >2+ or >500 mg | NA |
| Hematuria<br>(not to be reported<br>based on dipstick<br>findings or on blood<br>believed to be of<br>menstrual origin) | 6 to <10 RBCs per<br>high power field | ≥10 RBCs per high<br>power field | Gross, with or without<br>clots OR With RBC<br>casts OR Intervention<br>indicated | Life-threatening<br>consequences |
| Proteinuria<br>(random collection<br>tested by dipstick) | 1+ | 2+ | 3+ or higher | NA |

# ATTACHMENT 2: BLOOD PRESSURE LEVELS BY AGE AND HEIGHT PERCENTILES

# Blood Pressure Levels for Boys by Age and Height Percentile

| | ВР | | Systolic BP (mmHg) | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | ← Percentile of Height → | | | | | • | Perce | ntile of | Height | : → | | | |
| (Year) | • | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5t | 10th | 25th | 50th | 75th | 90th | 95th |
| 1 | 50th | 80 | 81 | 83 | 85 | 87 | 88 | 89 | 3 | 1 35 | 36 | 37 | 38 | 39 | 39 |
| | 90th | 94 | 95 | 97 | 99 | 100 | 102 | 103 | 4 | 9 50 | 51 | 52 | 53 | 53 | 54 |
| | 95th | 98 | 99 | 101 | 103 | 104 | 106 | 106 | 5 | 1 54 | 55 | 56 | 57 | 58 | 58 |
| | 99th | 105 | 106 | 108 | 110 | 112 | 113 | 114 | 6 | 1 62 | 63 | 64 | 65 | 66 | 66 |
| 2 | 50th | 84 | 85 | 87 | 88 | 90 | 92 | 92 | 3 | 9 40 | 41 | 42 | 43 | 44 | 44 |
| | 90th | 97 | 99 | 100 | 102 | 104 | 105 | 106 | 5 | 1 55 | 56 | 57 | 58 | 58 | 59 |
| | 95th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 5 | 9 59 | 60 | 61 | 62 | 63 | 63 |
| | 99th | 109 | 110 | 111 | 113 | 115 | 117 | 117 | 6 | 67 | 68 | 69 | 70 | 71 | 71 |
| 3 | 50th | 86 | 87 | 89 | 91 | 93 | 94 | 95 | 4 | 1 44 | 45 | 46 | 47 | 48 | 48 |
| | 90th | 100 | 101 | 103 | 105 | 107 | 108 | 109 | 5 | 9 59 | 60 | 61 | 62 | 63 | 63 |
| | 95th | 104 | 105 | 107 | 109 | 110 | 112 | 113 | 6 | 3 63 | 64 | 65 | 66 | 67 | 67 |
| | 99th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 7 | 1 71 | 72 | 73 | 74 | 75 | 75 |
| 4 | 50th | 88 | 89 | 91 | 93 | 95 | 96 | 97 | 4 | 7 48 | 49 | 50 | 51 | 51 | 52 |
| | 90th | 102 | 103 | 105 | 107 | 109 | 110 | 111 | 6 | 2 63 | 64 | 65 | 66 | 66 | 67 |
| | 95th | 106 | 107 | 109 | 111 | 112 | 114 | 115 | 6 | 67 | 68 | 69 | 70 | 71 | 71 |
| | 99th | 113 | 114 | 116 | 118 | 120 | 121 | 122 | 7 | 1 75 | 76 | 77 | 78 | 78 | 79 |
| 5 | 50th | 90 | 91 | 93 | 95 | 96 | 98 | 98 | 5 | 51 | 52 | 53 | 54 | 55 | 55 |
| | 90th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 6 | 5 66 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 108 | 109 | 110 | 112 | 114 | 115 | 116 | 6 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 99th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 7 | 7 78 | 79 | 80 | 81 | 81 | 82 |
| 6 | 50th | 91 | 92 | 94 | 96 | 98 | 99 | 100 | 5 | 3 53 | 54 | 55 | 56 | 57 | 57 |
| | 90th | 105 | 106 | 108 | 110 | 111 | 113 | 113 | 6 | 8 68 | 69 | 70 | 71 | 72 | 72 |
| | 95th | 109 | 110 | 112 | 114 | 115 | 117 | 117 | 7 | 2 72 | 73 | 74 | 75 | 76 | 76 |
| | 99th | 116 | 117 | 119 | 121 | 123 | 124 | 125 | 8 | 0 80 | 81 | 82 | 83 | 84 | 84 |
| 7 | 50th | 92 | 94 | 95 | 97 | 99 | 100 | 101 | 5 | 5 55 | 56 | 57 | 58 | 59 | 59 |
| | 90th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 7 | 70 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 110 | 111 | 113 | 115 | 117 | 118 | 119 | 7 | 1 74 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 8 | 2 82 | 83 | 84 | 85 | 86 | 86 |
| 8 | 50th | 94 | 95 | 97 | 99 | 100 | 102 | 102 | 5 | 5 57 | 58 | 59 | 60 | 60 | 61 |
| | 90th | 107 | 109 | 110 | 112 | 114 | 115 | 116 | 7 | 1 72 | 72 | 73 | 74 | 75 | 76 |
| | 95th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 7 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 99th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 8 | 84 | 85 | 86 | 87 | 87 | 88 |
| 9 | 50th | 95 | 96 | 98 | 100 | 102 | 103 | 104 | 5 | 7 58 | 59 | 60 | 61 | 61 | 62 |
| | 90th | 109 | 110 | 112 | 114 | 115 | 117 | 118 | 7 | 2 73 | 74 | 75 | 76 | 76 | 77 |
| | 95th | 113 | 114 | 116 | 118 | 119 | 121 | 121 | 7 | 3 77 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 120 | 121 | 123 | 125 | 127 | 128 | 129 | 8 | 1 85 | 86 | 87 | 88 | 88 | 89 |
| 10 | 50th | 97 | 98 | 100 | 102 | 103 | 105 | 106 | 5 | 3 59 | 60 | 61 | 61 | 62 | 63 |
| | 90th | 111 | 112 | 114 | 115 | 117 | 119 | 119 | 7 | 3 73 | 74 | 75 | 76 | 77 | 78 |
| | 95th | 115 | 116 | 117 | 119 | 121 | 122 | 123 | 7 | 7 78 | 79 | 80 | 81 | 81 | 82 |
| | 99th | 122 | 123 | 125 | 127 | 128 | 130 | 130 | 8 | 5 86 | 86 | 88 | 88 | 89 | 90 |

## Blood Pressure Levels for Boys by Age and Height Percentile (Continued)

| | ВР | | Systolic BP (mmHg) | | | | | | | Diastolic BP (mmHg) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | • | Perce | ntile of | Height | <b>→</b> | | | • | Perce | ntile of | Height | <b>→</b> | |
| (Year) | ullet | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 99 | 100 | 102 | 104 | 105 | 107 | 107 | 59 | 59 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 113 | 114 | 115 | 117 | 119 | 120 | 121 | 74 | 74 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 117 | 118 | 119 | 121 | 123 | 124 | 125 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 124 | 125 | 127 | 129 | 130 | 132 | 132 | 86 | 86 | 87 | 88 | 89 | 90 | 90 |
| 12 | 50th | 101 | 102 | 104 | 106 | 108 | 109 | 110 | 59 | 60 | 61 | 62 | 63 | 63 | 64 |
| | 90th | 115 | 116 | 118 | 120 | 121 | 123 | 123 | 74 | 75 | 75 | 76 | 77 | 78 | 79 |
| | 95th | 119 | 120 | 122 | 123 | 125 | 127 | 127 | 78 | 79 | 80 | 81 | 82 | 82 | 83 |
| | 99th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 86 | 87 | 88 | 89 | 90 | 90 | 91 |
| 13 | 50th | 104 | 105 | 106 | 108 | 110 | 111 | 112 | 60 | 60 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 117 | 118 | 120 | 122 | 124 | 125 | 126 | 75 | 75 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 124 | 126 | 128 | 129 | 130 | 79 | 79 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 130 | 131 | 133 | 135 | 136 | 137 | 87 | 87 | 88 | 89 | 90 | 91 | 91 |
| 14 | 50th | 106 | 107 | 109 | 111 | 113 | 114 | 115 | 60 | 61 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 120 | 121 | 123 | 125 | 126 | 128 | 128 | 75 | 76 | 77 | 78 | 79 | 79 | 80 |
| | 95th | 124 | 125 | 127 | 128 | 130 | 132 | 132 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 87 | 88 | 89 | 90 | 91 | 92 | 92 |
| 15 | 50th | 109 | 110 | 112 | 113 | 115 | 117 | 117 | 61 | 62 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 122 | 124 | 125 | 127 | 129 | 130 | 131 | 76 | 77 | 78 | 79 | 80 | 80 | 81 |
| | 95th | 126 | 127 | 129 | 131 | 133 | 134 | 135 | 81 | 81 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 134 | 135 | 136 | 138 | 140 | 142 | 142 | 88 | 89 | 90 | 91 | 92 | 93 | 93 |
| 16 | 50th | 111 | 112 | 114 | 116 | 118 | 119 | 120 | 63 | 63 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 125 | 126 | 128 | 130 | 131 | 133 | 134 | 78 | 78 | 79 | 80 | 81 | 82 | 82 |
| | 95th | 129 | 130 | 132 | 134 | 135 | 137 | 137 | 82 | 83 | 83 | 84 | 85 | 86 | 87 |
| | 99th | 136 | 137 | 139 | 141 | 143 | 144 | 145 | 90 | 90 | 91 | 92 | 93 | 94 | 94 |
| 17 | 50th | 114 | 115 | 116 | 118 | 120 | 121 | 122 | 65 | 66 | 66 | 67 | 68 | 69 | 70 |
| | 90th | 127 | 128 | 130 | 132 | 134 | 135 | 136 | 80 | 80 | 81 | 82 | 83 | 84 | 84 |
| | 95th | 131 | 132 | 134 | 136 | 138 | 139 | 140 | 84 | 85 | 86 | 87 | 87 | 88 | 89 |
| | 99th | 139 | 140 | 141 | 143 | 145 | 146 | 147 | 92 | 93 | 93 | 94 | 95 | 96 | 97 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for boys with height percentiles given in Table 3 (i.e., the 5th, 10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

 $<sup>^{*}</sup>$  The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

# Blood Pressure Levels for Girls by Age and Height Percentile

| | BP | | Systolic BP (mmHg) | | | | | | | Diasto | lic BP | mmHg | ) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | ← Percentile of Height → | | | | + | - Perce | ntile of | Height | <b>→</b> | | | | |
| (Year) | • | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 1 | 50th | 83 | 84 | 85 | 86 | 88 | 89 | 90 | 38 | 39 | 39 | 40 | 41 | 41 | 42 |
| | 90th | 97 | 97 | 98 | 100 | 101 | 102 | 103 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 95th | 100 | 101 | 102 | 104 | 105 | 106 | 107 | 56 | 57 | 57 | 58 | 59 | 59 | 60 |
| | 99th | 108 | 108 | 109 | 111 | 112 | 113 | 114 | 64 | 64 | 65 | 65 | 66 | 67 | 67 |
| 2 | 50th | 85 | 85 | 87 | 88 | 89 | 91 | 91 | 43 | 44 | 44 | 45 | 46 | 46 | 47 |
| | 90th | 98 | 99 | 100 | 101 | 103 | 104 | 105 | 57 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 95th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 99th | 109 | 110 | 111 | 112 | 114 | 115 | 116 | 69 | 69 | 70 | 70 | 71 | 72 | 72 |
| 3 | 50th | 86 | 87 | 88 | 89 | 91 | 92 | 93 | 47 | 48 | 48 | 49 | 50 | 50 | 51 |
| | 90th | 100 | 100 | 102 | 103 | 104 | 106 | 106 | 61 | 62 | 62 | 63 | 64 | 64 | 65 |
| | 95th | 104 | 104 | 105 | 107 | 108 | 109 | 110 | 65 | 66 | 66 | 67 | 68 | 68 | 69 |
| | 99th | 111 | 111 | 113 | 114 | 115 | 116 | 117 | 73 | 73 | 74 | 74 | 75 | 76 | 76 |
| 4 | 50th | 88 | 88 | 90 | 91 | 92 | 94 | 94 | 50 | 50 | 51 | 52 | 52 | 53 | 54 |
| | 90th | 101 | 102 | 103 | 104 | 106 | 107 | 108 | 64 | 64 | 65 | 66 | 67 | 67 | 68 |
| | 95th | 105 | 106 | 107 | 108 | 110 | 111 | 112 | 68 | 68 | 69 | 70 | 71 | 71 | 72 |
| | 99th | 112 | 113 | 114 | 115 | 117 | 118 | 119 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| 5 | 50th | 89 | 90 | 91 | 93 | 94 | 95 | 96 | 52 | 53 | 53 | 54 | 55 | 55 | 56 |
| | 90th | 103 | 103 | 105 | 106 | 107 | 109 | 109 | 66 | 67 | 67 | 68 | 69 | 69 | 70 |
| | 95th | 107 | 107 | 108 | 110 | 111 | 112 | 113 | 70 | 71 | 71 | 72 | 73 | 73 | 74 |
| | 99th | 114 | 114 | 116 | 117 | 118 | 120 | 120 | 78 | 78 | 79 | 79 | 80 | 81 | 81 |
| 6 | 50th | 91 | 92 | 93 | 94 | 96 | 97 | 98 | 54 | 54 | 55 | 56 | 56 | 57 | 58 |
| | 90th | 104 | 105 | 106 | 108 | 109 | 110 | 111 | 68 | 68 | 69 | 70 | 70 | 71 | 72 |
| | 95th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 72 | 72 | 73 | 74 | 74 | 75 | 76 |
| | 99th | 115 | 116 | 117 | 119 | 120 | 121 | 122 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| 7 | 50th | 93 | 93 | 95 | 96 | 97 | 99 | 99 | 55 | 56 | 56 | 57 | 58 | 58 | 59 |
| | 90th | 106 | 107 | 108 | 109 | 111 | 112 | 113 | 69 | 70 | 70 | 71 | 72 | 72 | 73 |
| | 95th | 110 | 111 | 112 | 113 | 115 | 116 | 116 | 73 | 74 | 74 | 75 | 76 | 76 | 77 |
| | 99th | 117 | 118 | 119 | 120 | 122 | 123 | 124 | 81 | 81 | 82 | 82 | 83 | 84 | 84 |
| 8 | 50th | 95 | 95 | 96 | 98 | 99 | 100 | 101 | 57 | 57 | 57 | 58 | 59 | 60 | 60 |
| | 90th | 108 | 109 | 110 | 111 | 113 | 114 | 114 | 71 | 71 | 71 | 72 | 73 | 74 | 74 |
| | 95th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 99th | 119 | 120 | 121 | 122 | 123 | 125 | 125 | 82 | 82 | 83 | 83 | 84 | 85 | 86 |
| 9 | 50th | 96 | 97 | 98 | 100 | 101 | 102 | 103 | 58 | 58 | 58 | 59 | 60 | 61 | 61 |
| | 90th | 110 | 110 | 112 | 113 | 114 | 116 | 116 | 72 | 72 | 72 | 73 | 74 | 75 | 75 |
| | 95th | 114 | 114 | 115 | 117 | 118 | 119 | 120 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 99th | 121 | 121 | 123 | 124 | 125 | 127 | 127 | 83 | 83 | 84 | 84 | 85 | 86 | 87 |
| 10 | 50th | 98 | 99 | 100 | 102 | 103 | 104 | 105 | 59 | 59 | 59 | 60 | 61 | 62 | 62 |
| | 90th | 112 | 112 | 114 | 115 | 116 | 118 | 118 | 73 | 73 | 73 | 74 | 75 | 76 | 76 |
| | 95th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 99th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 84 | 84 | 85 | 86 | 86 | 87 | 88 |

## Blood Pressure Levels for Girls by Age and Height Percentile (Continued)

| | BP | Systolic BP (mmHg) | | | | | | | Diastolic BP (mmHg) | | | | | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Age | Percentile | | + | Perce | ntile of | Height | <b>→</b> | | | + | Perce | ntile of | Height | <b>→</b> | |
| (Year) | • | 5th | 10th | 25th | 50th | 75th | 90th | 95th | 5th | 10th | 25th | 50th | 75th | 90th | 95th |
| 11 | 50th | 100 | 101 | 102 | 103 | 105 | 106 | 107 | 60 | 60 | 60 | 61 | 62 | 63 | 63 |
| | 90th | 114 | 114 | 116 | 117 | 118 | 119 | 120 | 74 | 74 | 74 | 75 | 76 | 77 | 77 |
| | 95th | 118 | 118 | 119 | 121 | 122 | 123 | 124 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 99th | 125 | 125 | 126 | 128 | 129 | 130 | 131 | 85 | 85 | 86 | 87 | 87 | 88 | 89 |
| 12 | 50th | 102 | 103 | 104 | 105 | 107 | 108 | 109 | 61 | 61 | 61 | 62 | 63 | 64 | 64 |
| | 90th | 116 | 116 | 117 | 119 | 120 | 121 | 122 | 75 | 75 | 75 | 76 | 77 | 78 | 78 |
| | 95th | 119 | 120 | 121 | 123 | 124 | 125 | 126 | 79 | 79 | 79 | 80 | 81 | 82 | 82 |
| | 99th | 127 | 127 | 128 | 130 | 131 | 132 | 133 | 86 | 86 | 87 | 88 | 88 | 89 | 90 |
| 13 | 50th | 104 | 105 | 106 | 107 | 109 | 110 | 110 | 62 | 62 | 62 | 63 | 64 | 65 | 65 |
| | 90th | 117 | 118 | 119 | 121 | 122 | 123 | 124 | 76 | 76 | 76 | 77 | 78 | 79 | 79 |
| | 95th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 80 | 80 | 80 | 81 | 82 | 83 | 83 |
| | 99th | 128 | 129 | 130 | 132 | 133 | 134 | 135 | 87 | 87 | 88 | 89 | 89 | 90 | 91 |
| 14 | 50th | 106 | 106 | 107 | 109 | 110 | 111 | 112 | 63 | 63 | 63 | 64 | 65 | 66 | 66 |
| | 90th | 119 | 120 | 121 | 122 | 124 | 125 | 125 | 77 | 77 | 77 | 78 | 79 | 80 | 80 |
| | 95th | 123 | 123 | 125 | 126 | 127 | 129 | 129 | 81 | 81 | 81 | 82 | 83 | 84 | 84 |
| | 99th | 130 | 131 | 132 | 133 | 135 | 136 | 136 | 88 | 88 | 89 | 90 | 90 | 91 | 92 |
| 15 | 50th | 107 | 108 | 109 | 110 | 111 | 113 | 113 | 64 | 64 | 64 | 65 | 66 | 67 | 67 |
| | 90th | 120 | 121 | 122 | 123 | 125 | 126 | 127 | 78 | 78 | 78 | 79 | 80 | 81 | 81 |
| | 95th | 124 | 125 | 126 | 127 | 129 | 130 | 131 | 82 | 82 | 82 | 83 | 84 | 85 | 85 |
| | 99th | 131 | 132 | 133 | 134 | 136 | 137 | 138 | 89 | 89 | 90 | 91 | 91 | 92 | 93 |
| 16 | 50th | 108 | 108 | 110 | 111 | 112 | 114 | 114 | 64 | 64 | 65 | 66 | 66 | 67 | 68 |
| | 90th | 121 | 122 | 123 | 124 | 126 | 127 | 128 | 78 | 78 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 128 | 130 | 131 | 132 | 82 | 82 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 132 | 133 | 134 | 135 | 137 | 138 | 139 | 90 | 90 | 90 | 91 | 92 | 93 | 93 |
| 17 | 50th | 108 | 109 | 110 | 111 | 113 | 114 | 115 | 64 | 65 | 65 | 66 | 67 | 67 | 68 |
| | 90th | 122 | 122 | 123 | 125 | 126 | 127 | 128 | 78 | 79 | 79 | 80 | 81 | 81 | 82 |
| | 95th | 125 | 126 | 127 | 129 | 130 | 131 | 132 | 82 | 83 | 83 | 84 | 85 | 85 | 86 |
| | 99th | 133 | 133 | 134 | 136 | 137 | 138 | 139 | 90 | 90 | 91 | 91 | 92 | 93 | 93 |

BP, blood pressure

For research purposes, the standard deviations in Appendix Table B–1 allow one to compute BP Z-scores and percentiles for girls with height percentiles given in Table 4 (i.e., the 5th, 10th, 25th, 50th, 75th, 90th, and 95th percentiles). These height percentiles must be converted to height Z-scores given by (5% = -1.645; 10% = -1.28; 25% = -0.68; 50% = 0; 75% = 0.68; 90% = 1.28%; 95% = 1.645) and then computed according to the methodology in steps 2–4 described in Appendix B. For children with height percentiles other than these, follow steps 1–4 as described in Appendix B.

<sup>\*</sup> The 90th percentile is 1.28 SD, 95th percentile is 1.645 SD, and the 99th percentile is 2.326 SD over the mean.

# ATTACHMENT 3: STAGE-3-DEFINING OPPORTUNISTIC ILLNESSES IN HIV INFECTION

Bacterial infections, multiple or recurrent\*

Candidiasis of bronchi, trachea, or lungs

Candidiasis of esophagus

Cervical cancer, invasive<sup>†</sup>

Coccidioidomycosis, disseminated or extrapulmonary

Cryptococcosis, extrapulmonary

Cryptosporidiosis, chronic intestinal (>1 month's duration)

Cytomegalovirus disease (other than liver, spleen, or nodes), onset at age >1 month

Cytomegalovirus retinitis (with loss of vision)

Encephalopathy attributed to HIV§

Herpes simplex: chronic ulcers (>1 month's duration) or bronchitis, pneumonitis, or esophagitis (onset at age >1 month)

Histoplasmosis, disseminated or extrapulmonary

Isosporiasis, chronic intestinal (>1 month's duration)

Kaposi sarcoma

Lymphoma, Burkitt (or equivalent term)

Lymphoma, immunoblastic (or equivalent term)

Lymphoma, primary, of brain

Mycobacterium avium complex or Mycobacterium kansasii, disseminated or extrapulmonary

Mycobacterium tuberculosis of any site, pulmonary<sup>†</sup>, disseminated, or extrapulmonary

Mycobacterium, other species or unidentified species, disseminated or extrapulmonary

Pneumocystis jirovecii (previously known as "Pneumocystis carinii") pneumonia

Pneumonia, recurrent<sup>†</sup>

Progressive multifocal leukoencephalopathy

Salmonella septicemia, recurrent

Toxoplasmosis of brain, onset at age >1 month

Wasting syndrome attributed to HIV§

38

<sup>\*</sup> Only among children aged <6 years.

<sup>&</sup>lt;sup>†</sup> Only among adults, adolescents, and children aged ≥6 years.

<sup>§</sup> Suggested diagnostic criteria for these illnesses, which might be particularly important for HIV encephalopathy and HIV wasting syndrome, are described in the following references:

CDC. 1994 Revised classification system for human immunodeficiency virus infection in children less than 13 years of age. MMWR 1994;43(No. RR-12).

CDC. 1993 Revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. MMWR 1992;41(No. RR-17).

# **Signature**

| User | Date Reason |
|------|-------------|
|------|-------------|